CLINICAL TRIAL: NCT04253639
Title: Identification of Predictive Factors for observAnce of Transcutaneous Electrical NeuroStimulation (TENS) in Chronic Pain
Acronym: IPATENS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sublimed (Industry)
Responsible Party: Sponsor
Other Study IDs: IPATENS
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain
Keywords: TENS; Predictive factors; Compliance; Chronic pain
MeSH Terms: conditions — Chronic Pain; Patient Compliance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients must fill questionnaires to collect socio-demographics, aetiology and characteristics of pain, efficacy and tolerance regarding the TENS.
  Study sites must fill questionnaires to collect information regarding the type of pain management centre, the characteristics of the clinician, the characteristics of the TENS prescribed.

SUMMARY:
This is a retrospective and transverse multicenter study to identify predictive factors for adherence to TENS by chronic pain patients followed in structures specialized in Chronic Pain management (SPC).

The study contains 2 parts:

* A retrospective part of data collection in the patient follow-up file of the SPC during the 6 months elapsed after the first rental prescription.
* A transversal part, aimed at collecting additional information on the use of TENS, satisfaction and quality of life during a telephone interview after 6 months of use.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over when TENS was implemented.
* Suffering from chronic pain.
* Follow-up in nurse consultation within a centre specialized in chronic pain management identified and labeled by a local regulatory agency.
* Benefiting from the implementation of TENS for more than 6 months by a nurse from a centre specialized in chronic pain management.
* Affiliate or Beneficiary of a health insurance scheme.
* For patients in the study population: Having expressed their non-opposition to participate in the study.
* Patient used to verify the representativeness of the population studied: Unable to be contacted by phone and not having expressed their refusal to participate or for which the mail has not returned undelivered

Non-inclusion criteria

* Minor.
* Major incapable to oppose to the use of their data during the study due to medical or legal decision.
* Having language impairment.
* Having difficulties understanding the French language.
* Unable to participate in the phone survey.
* Not affiliated with Health Insurance / Social Security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied is all adult chronic pain patients, who have benefited from an initiation of treatment with TENS dating back at least 6 months within a centre specialized in chronic pain management identified and labeled by a local regulatory agency.
  Patients who agree to participate in the study will be recruited in reverse chronological order from the list of patients in the active queue of each centre. Ten patients will be recruited by each investigator with a total of 50 centers.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Determination of predictive factors explaining compliance to TENS. | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient
  Compliance is evaluated on a 6 month period prior to the inclusion. Compliant patients to TENS are defined as having 0, 1 or 2 to score of Morisky Medication Adherence Scale. Factors which can explain the lack of compliance will be collected and categorized within "pain centre", "clinician", "TENS characteristics", "patient socio-demographics", "aetiology and characteristics of pain", "efficacy and tolerance" data.

SECONDARY OUTCOMES:
Efficacy parameters: follow up visits | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: T1month, T3month, T6month
  Efficacy parameters: Rate of patients followed at 1, 3 and 6 months after the initiation session to TENS and rate and time of premature discontinuation of treatment.
Efficacy parameters: observance | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: T1month, T3month, T6month
  Rate of observant patients at 1, 3 and 6 months after the TENS initiation session.
Efficacy parameters: pain intensity | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: TENS initiation, T1month, T3month, T6month and on a 8-day period preceding the last use of TENS
  Pain intensity (PI) collected using an 11 point digital scale (EN) (0 - 10, 0 = no pain; 10 = maximum pain imaginable) during the first contact with the investigator/nurse (D0) (patient record), then 1, 3 and 6 months after the TENS initiation session (patient record) and during the 8 days preceding the last use of TENS.
Efficacy parameters: Pain intensity differences | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: TENS initiation, T1month, T3month, T6month and on a 8-day period preceding the last use of TENS
  Pain intensity differences (PID) on the average intensity scores at 1, 3 and 6 months after the TENS initiation session and during the 8 days preceding the last use of TENS (PI inclusion - PI T-time).
Efficacy parameters: Sum of Pain intensity differences | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: TENS initiation, T1month, T3month, T6month and on a 8-day period preceding the last use of TENS
  Sum of pain intensity differences (SPID) on the average intensity scores at 1, 3 and 6 months after the TENS initiation session and during the 8 days preceding the last use of TENS, weighted on the time factor: SPID0-Xmonth = Σ [T (i) -T (i-1)] xPID (i).
Efficacy parameters: punctual relief | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: TENS initiation, T1month, T3month, T6month and on a 8-day period preceding the last use of TENS
  Relief (PAR) using an 11-point numeric scale (0% -100%, 0 = no relief; 100% = complete relief) at 1, 3 and 6 months (patient record) after the introduction to TENS and during the 8 days preceding the last use of TENS.
Efficacy parameters: Total relief | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: TENS initiation, T1month, T3month, T6month and on a 8-day period preceding the last use of TENS
  Total relief (TOTPAR) or TOTPARt0-tx = Σ [T (x) -T (x-1)] xPAR (x) when T (0) = 0, T (x) is the selected evaluation time and PAR (x) is the PAR value at the times 1, 3 and 6 months after the TENS initiation session and during the 8 days preceding the last use of the TENS
Efficacy parameters: Quality of life | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: on the day of the last use of TENS
  Quality of life questionnaire (EQ-5D) when TENS was last used.
Efficacy parameters: Impression of change | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: on the day of the last use of TENS
  Patients' Global Impression of Change (PGIC) when the TENS was last used.
Efficacy parameters: Satisfaction | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient at the following timepoints: on the day of the last use of TENS
  Satisfaction when TENS was last used.
Efficacy parameters: wish for continuation | Data are collected the day of the inclusion.
  Number of patients wishing to continue treatment and purchase the device
Mode of use of the TENS | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient.
  For each of the 4 TENS allowed in the study, description of the program used and collection of the duration of use, the number of sessions per day and the duration of the post-effect as well as compliance with the instructions for use of the TENS during follow-up.
Tolerance parameters: AEs | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient.
  Number, delay of onset and type of serious and non-serious AEs (SAEs) occurring during the 6 months of follow-up and attributable, according to the opinion of the investigator, to treatment.
Tolerance parameters: premature discontinuation | Data are collected the day of the inclusion retrospectively on a 6 month period prior to the inclusion of each patient.
  Number of premature discontinuations before 6 months for tolerance problems

CONTACTS AND LOCATIONS:
Overall Officials: Muriel PERRIOT MOREY, Principal Investigator — Chateauroux hospital - Pain managment center

IPD SHARING:
Plan to Share IPD: No